CLINICAL TRIAL: NCT02063581
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Formulation on the Bioavailability of Ipatasertib (GDC-0068) in Healthy Subjects
Brief Title: A Study Evaluating the Effect of Formulation on the Bioavailability of Ipatasertib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP29066
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — ipatasertib; Capsules; Tablets

ARMS (2):
- Sequence 1: Tablet followed by Capsule (Experimental)
  Interventions: Drug: ipatasertib (Capsule); Drug: ipatasertib (Tablet)
- Sequence 2: Capsule followed by Tablet (Experimental)
  Interventions: Drug: ipatasertib (Capsule); Drug: ipatasertib (Tablet)

INTERVENTIONS:
Drug: ipatasertib (Capsule) — Orally administered single dose of Ipatasertib formulated as a capsule.
Drug: ipatasertib (Tablet) — Orally administered single dose of Ipatasertib formulated as a tablet.

SUMMARY:
This Phase I, open-label, randomized, 2-period crossover study was designed to determine the relative bioavailability of ipatasertib administered as capsule and tablet formulations to healthy adult volunteers. Participants will be randomized to one of two treatment sequences to receive a single oral administration of ipatasertib in tablet or capsule formulation followed, after a washout period, by a single oral administration of ipatasertib in the second formulation. Pharmacokinetics will be assessed, and standard physical and clinical evaluations will be performed throughout the study. Time on study is expected to be 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged 18 to 55 years, inclusive
* Body mass index (BMI) from 18.5-29.9 kg/m2, inclusive

Exclusion Criteria:

* Clinically significant findings from medical history or screening evaluations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve (AUC) of ipatasertib | Days 1-13
Maximum concentration (Cmax) reached of ipatasertib | Days 1-13
Time to maximum concentration (Tmax) of ipatasertib | Days 1-13

SECONDARY OUTCOMES:
Incidence of adverse events | From check-in (Day -1) to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Madison, Wisconsin, United States